CLINICAL TRIAL: NCT02702544
Title: Effect of Passive Leg Rasing on Changes in Volumetric Hemodynamic Parameters Induced by Fluid Removal
Brief Title: Effect of Passive Leg Raising for Fluid Responsiveness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 02.014.1MR
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Body Fluid Retention; Impedance; Cardiac Output, Low
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- neutral position (Experimental): the patient is in the neutral position, located on his back on a flat surface
  Interventions: Device: CardioScreen 1000 - Haemodynamic Measurement System, Medis; Device: SCHILLER, BR-102 plus - Ambulatory Blood Pressure Monitoring System
- legs raised for 20 degrees (Experimental): patient is placed on a flat surface, legs raised for 20 degrees, supported around ankles
  Interventions: Device: CardioScreen 1000 - Haemodynamic Measurement System, Medis; Device: SCHILLER, BR-102 plus - Ambulatory Blood Pressure Monitoring System
- legs raised for 30 degrees (Experimental): patient is placed on a flat surface, legs raised for 30 degrees, supported around ankles
  Interventions: Device: CardioScreen 1000 - Haemodynamic Measurement System, Medis; Device: SCHILLER, BR-102 plus - Ambulatory Blood Pressure Monitoring System
- legs raised for 45 degrees (Experimental): patient is placed on a flat surface, legs raised for 45 degrees, supported around ankles
  Interventions: Device: CardioScreen 1000 - Haemodynamic Measurement System, Medis; Device: SCHILLER, BR-102 plus - Ambulatory Blood Pressure Monitoring System
- legs raised for 60 degrees (Experimental): patient is placed on a flat surface, legs raised for 60 degrees, supported around ankles
  Interventions: Device: CardioScreen 1000 - Haemodynamic Measurement System, Medis; Device: SCHILLER, BR-102 plus - Ambulatory Blood Pressure Monitoring System

INTERVENTIONS:
Device: CardioScreen 1000 - Haemodynamic Measurement System, Medis — Impedance cardiography (ICG)
Device: SCHILLER, BR-102 plus - Ambulatory Blood Pressure Monitoring System — Blood pressure monitoring every 1 min during leg elevation

SUMMARY:
Changes in volumetric hemodynamic parameters and fluid overload (Cardiac Index,Stroke Volume, Thoracic Fluid Content, Systemic Vascular Resistance) were measured using a impedance cardiography (ICG) (CardioScreen 1000 - Haemodynamic Measurement System, Medis. GmbH Ilmenau) while lifting the leg at different angles. The measurement lasted 12 minutes.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* no clinical cardiovascular disease during the 6 months proceeding entry

Exclusion Criteria:

* not meet above criteria
* episode of illness (for example: infection)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Changes in volumetric hemodynamic parameter- cardiac index [l/min/m2]) induced by fluid removal on leg elevation | 1 day

SECONDARY OUTCOMES:
Changes in volumetric hemodynamic parameter- stroke volume [ml] induced by fluid removal on leg elevation | 1 day
Changes in volumetric hemodynamic parameter- systemic vascular resistance index [dyn·s·cm-5·m-2] induced by fluid removal on leg elevation | 1 day
Changes in fluid removal parameter- thoracic fluid content [1/kOhm] during leg elevation | 1 day
Changes in blood pressure values [mmHg] induced by fluid removal on leg elevation | 1 day
Changes in vascular parameter- thoracic arterial complicance [ml/mmHg/m-2] during leg elevation | 1 day
Changes in contractility parameter- acceleration index [1/100/s-2] during leg elevation | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Department of Emergency Medicine, Warsaw, Masovia, Poland